CLINICAL TRIAL: NCT06745765
Title: Effects of Virtual Reality in the Management of Anxiety in Patients Undergoing Interventional Radiology Procedures: Randomized Study
Brief Title: Virtual Reality for Anxiety in Interventional Radiology Procedures
Acronym: VR-IR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Giancarlo Facchini, Medical Doctor, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CE AVEC: 622/2024/Sper/IOR
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Preoperative Anxiety
Keywords: Virtual reality; Preoperative care

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR (Experimental): Patients will use virtual reality before the procedure in addition to usual preoperative care.
  Interventions: Device: Virtual reality headset
- NO VR (No Intervention): Patients will not use virtual reality; hence, they will experience usual preoperative care.

INTERVENTIONS:
Device: Virtual reality headset — Patients will use virtual reality before the procedure in addition to usual preoperative care.
  Arms: VR

SUMMARY:
The goal of this clinical trial is to learn if virtual reality works to reduce anxiety in patients undergoing interventional radiology procedures. The main questions it aims to answer are:

Does virtual reality lower anxiety in patients undegoing minimally invasive procedures? Can it help the platient's compliance and operators' satisfaction? Researchers will compare virtual reality to usual preoperative care to see if virtual reality is effective.

Participants will:

Use virtual reality for 20 minutes before the intervention starts. Complete questionnaires before and after the procedure.

DETAILED DESCRIPTION:
Patients enrolled and assigned to group 1 will wear the virtual reality visor in the induction room, before entering the Angio Suite in which the procedure will take place. The study requires that before and at the end of the procedure, a measurement of blood pressure and heart rate in order to measure the change in the patient's anxiety state. At the end of the procedure, they will be administered satisfaction tests to interventional radiologists and patients. The viewers in question are Meta Quest 2. Through the use of these viewers, the patient will will watch a VR video containing music and natural images that can promote relaxation in preparation for the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Indication to CT-guided biopsy in local anesthesia
* Informed consent signature

Exclusion Criteria:

* Lack of patient consent to trial.
* Lack of eligibility to perform CT-guided needle biopsy, or eligibility to perform the procedure but with administration of general anesthesia or sedation.
* patients who do not speak Italian or English will be excluded;
* patients with visual and/or hearing impairment;
* patients on analgesics or anxiolytics;
* patients with the following conditions: dementia, psychiatric disorders; headache, dizziness, recent head injury, epilepsy, and other conditions in which the application of VR glasses has been judged to be potentially harmful; and when the topical anesthetic (lidocaine and prilocaine [eutectic mixture of local anesthetic (EMLA)]) or tetracaine (Ametop) was not properly applied before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety change in STAI-S scale | At baseline (before VR), after 15 minutes, after 1 hour
  This subscale measures state anxiety, which is the anxiety temporary that an individual experiences in a specific situation. È designed to assess an individual's reaction to a particular event or situation particular moment at a specific time. Questions are phrased to reflect feelings such as tension, worry, agitation, and nervousness. Each item is formulated as a statement to which individuals must respond by indicating their level of agreement or discomfort on a 4-point scale.
  Scoring system:
  * 20-37: Low Anxiety
  * 38-44: Moderate anxiety
  * 45-80: High anxiety A difference of at least 3 points on the scale between the two groups is considered significant.
  Scores will be assessed before and after the use of virtual reality (for patients in VR group) and after the procedure.

SECONDARY OUTCOMES:
Change of anxiety (VAS-A score) | At baseline (before VR), after 15 minutes, after 1 hour
  The VAS-A scale, short for "Visual Analogue Scale for Anxiety," is an instrument used in the subjective assessment of anxiety. It consists of a horizontal line usually about 10 centimeters long, with ends marked by two descriptions opposites related to the degree of perceived anxiety. For example, one end may be labeled "no anxiety" and on the other "extreme anxiety." Scores will be assessed before and after the use of virtual reality (for patients in VR group) and after the procedure.
Change in heart rate | At baseline (before VR), after 15 minutes, after 1 hour
  Heart rate will be measured before and after the use of virtual reality (for patients in the Vr group) and after the procedure. Heart rate may exceed 100 bpm during an anxiety episode (range of normal at rest 60-100 bpm).
Change in blood pressure | At baseline (before VR), after 15 minutes, after 1 hour
  An anxious state will be considered as an increase in pressure relative to normal (generally considered to be around 120/80 mmHg), thus, indicatively, values of 140/90 mmHg or more.
  Blood pressure will be measured before and after the use of virtual reality (for patients in VR group) and after the procedure.
Patient satisfaction on a scale from 0 to 10 | After 1 hour
  0=totally unsatisfied 10= totally satisfied
Operator satisfaction on a 0-10 scale | After 1 hour
  0 = totally unsatisfied with patient's compliance 10 = totally satisfied with patient's compliance

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns.